CLINICAL TRIAL: NCT03213756
Title: Effect of Isometric Preoperative Exercise on Vascular Caliber and the Maturation of Autologous Arteriovenous Fistulas. Randomized Clinical Trial
Brief Title: Isometric Preoperative Exercise on Autologous Arteriovenous Fistulas. Randomized Clinical Trial
Acronym: PHYSICALFAV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Collaborators: Spanish Society of Nephrology (Other)
Responsible Party: Principal Investigator, Ines Aragoncillo, Nephrologist, Hospital General Universitario Gregorio Marañon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHYSICALFAV; PHYSICALFAV (Other: CEIC COMUNIDAD AUTÓNOMA MADRID (24.05.17)); PHYSICALFAV (Other: CEIC HOSPITAL GREGORIO MARAÑON (29.6.17))
Record Dates: First submitted 2017-06-29; First posted 2017-07-11 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Arteriovenous Fistula Thrombosis; Arteriovenous Fistula Stenosis
Keywords: doppler ultrasound; physical exercise; arteriovenous fistula maturation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Open-label, prospective, controlled, randomized, multicenter study in parallel groups, where in the preoperative AVF period, one group of patients will perform an isometric exercise protocol for 8 weeks and will be compared with a control group of patients that will not perform this preoperative exercise
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative isometric exercise (PIE) group (Experimental): In the PIE group, the patients will perform daily preoperative exercise protocol based on isometric exercises using hand grip and elastic bands. They will perform this protocol for at least six and ideally eight weeks before surgery.
  Interventions: Device: Isometric exercises using Hand grip and elastic bands
- Control group (No Intervention): Control group patients will follow the usual surgical waiting list protocol (Estimated 1,5-2 months).

INTERVENTIONS:
Device: Isometric exercises using Hand grip and elastic bands — * Isometric exercises using hand-grip. This exercise consists of two sets of 30 hand-grip contractions with the hand of the upper arm candidate for AVF (in case of doubts about the most appropriate arm for AVF the exercise will be performed with both arms). The patient will rest one minute every 10 contractions and 5 minutes between both sets. The patient will repeat this protocol twice a day, morning and night (Approximately 15 minutes each session). The contraction intensity will start with half of the maximum force obtained by dynamometry and will be increased or decreased to be placed on an effort intensity 2-3 in the Borg scale.
  * Isometric exercise using elastic bands. At noon the patient will perform a slow contraction session using elastic band with 20 slow repetitions with the arm in flexion and 20 repetitions with the arm in extension. (Total duration: less than 10 minutes)
  Arms: Preoperative isometric exercise (PIE) group

SUMMARY:
A good vascular access (VA) is vital for hemodialysis (HD) patients. The start of HD with autologous arteriovenous fistula (AVF) means higher survival, lower sanitary costs and complications. The distal forearm AVF is known as the best option but not all patients are good candidates for this surgery, and there is a primary failure rate between 20 and 50% published in literature.

The choice of the optimal AVF for each patient is conditioned mainly by the anatomical and hemodynamic characteristics of the artery and the vein chosen to perform the anastomosis. These characteristics can be modified by performing physical exercise Some vascular access guidelines suggest the performance of isometric exercises in the pre and postoperative period of the AVF confection. However, there is very little data in literature on the possible efficacy of preoperative exercise, although small published observational studies point to an improvement in the venous and arterial caliber. Regarding the postoperative exercises, they do seem to improve maturation, however the degree of evidence in literature is low and there is no consensus on the exercise protocol to follow.

We present an open-label, multicenter, prospective, controlled and randomized study in order to evaluate the usefulness of preoperative isometric exercise (PIE) in pre-dialysis patients or in prevalent HD with indication of performing a new AVF. The randomization will be 1: 1, one group of patients will perform PIE for 8 weeks and the other group of patients will be a control group. The main purpose will be to evaluate if there is a lower rate of primary failure in the PIE group compared with control group.

DETAILED DESCRIPTION:
RECRUITING PERIOD: 20 months.

FOLLOW UP: From the first preoperative assessment visit for AVF up to 3 months after its creation.

METHODS:

After signing the informed consent, patients will be randomized through a centralized computer program to one of two groups of patients, PIE group versus control group.

In both groups of patients, a first physical examination of upper arm extremities and an initial doppler ultrasound will be performed, evaluating the anatomical and hemodynamic characteristics of the arteries and veins of both arms. At that time, a first surgical option of AVF will be indicated.

In the PIE group, the patients will receive detailed information about the daily preoperative exercise protocol and they will perform this protocol for at least six and ideally more than eight weeks based on:

* Isometric exercise using hand-grip. This exercise consists of two sets of 30 hand-grip contractions with the hand of the upper arm candidate for AVF (in case of doubts about the most appropriate arm for AVF the exercise will be performed with both arms). The patient will rest one minute every 10 contractions and 5 minutes between both sets. The patient will repeat this protocol twice a day, morning and night (Approximately 15 minutes each session). The contraction intensity will start with half of the maximum force obtained by dynamometry and will be increased or decreased to be placed on an effort intensity 2-3 in the Borg scale.
* Isometric exercise using elastic bands. At noon the patient will perform a slow contraction session using elastic band with 20 slow repetitions with the arm in flexion and 20 repetitions with the arm in extension. (Total duration: less than 10 minutes) Clinical follow-up of these patients will be fortnightly to ensure that they perform the exercises correctly and to measure the force acquired through dynamometry. Likewise, brachial diameter and bicipital and tricipital skinfolds will be measured. In addition, they will be contacted by telephone once a week to assess compliance. Doppler ultrasonography will be performed at the initial visit, and at 4 and 8 week-visits (visits 1, 2 and 3). In the doppler ultrasound performed at 8 weeks, the final surgical indication will be given depending on the caliber of the vessels in the chosen arm. At the initial visit and at the 8-week visit, biological samples will be obtained to assess the parameters of nutrition and muscle mass and a bioimpedanciometry will be performed.

The date of surgery will be coordinated with anesthesia and peripheral vascular surgery services to program the intervention during the fortnight after the 8-week isometric exercise period (weeks 9-10). In prevalent HD patients with central venous catheter (CVC) presenting greater urgency of AVF, surgery will be scheduled between the 6 and 8 week of exercises.

Control group patients will follow the usual surgical waiting list protocol (Estimated 1,5-2 months). Baseline and preoperative ultrasonography will also be performed in these patients, in which it will be verified that there are no significant changes in vascular mapping (punctures sites, hematomas, etc.) and the indication of AVF performed in the initial visit will be confirmed. Dynamometry, bicipital and tricipital skinfolds measurement, brachial diameter, analytical parameters of nutrition and muscle mass and bioimpedanciometry will be performed both at the onset visit and at the preoperative visit. The only difference with PIE group is the 4 weeks follow-up ultrasound that will not be performed in control group.

After the AVF creation the maturation will be monitored with doppler ultrasound at 1, 6 and 12 weeks after the surgery (visits 4, 5 and 6) and the usual postoperative isometric exercise with ball contraction will be recommended to all patients. Follow-up will be completed three months after the surgical procedure, defining whether the AVF has matured or if there has been a primary failure.

FOLLOW-UP LOSSES:

* Abandonment or withdrawal of informed consent.
* Transplant.
* Change of dialysis technique.
* Transfer to another center.
* Exitus.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signature.
* Age between 18 and 89 years.
* Patients with advanced chronic kidney disease, stages IV-V, in pre-dialysis or prevalent HD patients, requiring new AVF.

Exclusion Criteria:

* Absence of adequate arteries and veins to allow autologous AVF. (The minimum gauges that will be considered in order to perform an autologous AVF are: artery caliber equal or greater than 1.6 mm and vein caliber equal or greater than 1,8 mm with a compressor).
* Diagnosis of coagulopathy or hemoglobinopathy of any cause.
* Patients who urgently need an AVF without the possibility of being 8 weeks on the surgical waiting list.
* Impossibility to perform the physical exercise protocol due to physical or mental disabilities or lack of social support.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Impact of PIE on AVF primary failure comparing the control group and the PIE group. | 12 weeks after AVF surgery (visit 6)
  We will evaluate in both groups the primary failure rate. It will be evaluated during visit 6 (12 weeks after AVF creation). We expect a lower primary failure rate in the PIE group.

SECONDARY OUTCOMES:
Percentage of candidate patients for autologous distal or proximal AVF in both groups. | 1 week after AVF surgery (visit 4)
  We will evaluate how many distal or proximal AVFs we perform in both groups. We expect an increase in the percentage of distal AVF in the PIE group
Differences on the caliber of upper arm arteries and veins in the PIE group before and after isometric exercise. | 8 weeks follow up visit before surgery (visit 3)
  Caliber, resistance index and flow of radial and brachial arteries and caliber of cephalic and basilic veins wil be measured in both groups using doppler ultrasound. We expect to find an increase in the diameters of arteries and veins in PIE group.
Impact of AVF evaluation with doppler ultrasound in the postoperative period in both groups, adding the usual isometric exercise with ball contraction in all patients. | 12 weeks after AVF surgery (visit 6)
  This study will allow to protocolize the AVF maturation surveillance with Doppler ultrasound in all participating centers, with early detection of stenosis and optimization of the primary assisted patency of AVF in our patients.
Analysis of the optimal arterial and venous calibres to minimize the primary failure of AVF according to the individual risk factors in both groups of patients. | 12 weeks after AVF surgery (visit 6)
  We will correlate the characteristics of arteria and vein and comorbidities of the patients with the AVFs outcomes in both groups in order to find the optimal characteristics of arteria and vein to perform an adequate AVF
Impact of nutritional-inflammatory status on AVF outcomes | 12 weeks after AVF surgery (visit 6)
  We will study if there is any correlation between nutritional-inflammatory status of the patients included in both groups and the AVF outcomes.
  The nutritional-inflammatory status will be evaluated with clinical and biochemical parameters, including endothelial disfunction biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: INES ARAGONCILLO, MD, Principal Investigator — GREGORIO MARAÑON HOSPITAL; ALMUDENA VEGA, MD PHD, Study Chair — GREGORIO MARAÑON HOSPITAL; SORAYA ABAD, MD, Study Chair — GREGORIO MARAÑON HOSPITAL; NICOLAS MACIAS, MD, Study Chair — GREGORIO MARAÑON HOSPITAL; JOSE MANUEL LIGERO, MD, Study Chair — GREGORIO MARAÑON HOSPITAL; ROSARIO GARCIA PAJARES, MD, Study Chair — GREGORIO MARAÑON HOSPITAL; ANGEL LUIS MORALES, MD, Study Chair — GREGORIO MARAÑON HOSPITAL; TERESA CERVERA, MD, Study Chair — GREGORIO MARAÑON HOSPITAL; JAVIER RIO, MD, Study Chair — GREGORIO MARAÑON HOSPITAL; DIEGO RUIZ CHIRIBOGA, MD, Study Chair — GREGORIO MARAÑON HOSPITAL; ELENA MENENDEZ, MD, Study Chair — GREGORIO MARAÑON HOSPITAL; MARTA ALBALATE, MD PHD, Study Chair — HOSPITAL INFANTA LEONOR; JARA AMPUERO, MD, Study Chair — HOSPITAL DEL SURESTE; COVADONGA HEVIA, MD, Study Chair — Hospital Infanta Sofia; SILVIA CALDES, MD, Study Chair — Hospital Infanta Sofia; YESIKA AMEZQUITA, MD, Study Chair — Hospital Infanta Sofia; YOLANDA HERNANDEZ, MD, Study Chair — Hospital Infanta Sofia; CRISTINA MORATILLA, MD PHD, Study Chair — CLINICA FUENSANTA; CARMEN CABRE, MD, Study Chair — CLINICA FUENSANTA; JOSE LUIS MARTIN CONTY, Study Chair — CASTILLA LA MANCHA UNIVERSITY; CRISTINA FERNANDEZ, MD PHD, Study Chair — Hospital Clinico de Madrid; ISRAEL LEBLIC, MD, Study Chair — Hospital Universitario La Paz
Locations (1):
- Hospital Gregorio Marañon, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Primary and secondary outcome results will be included in the web site with in 12 month from the end of the study
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Primary and secondary outcome results will be included in the web site with in 12 month from the end of the study
Access Criteria: Public access
URL: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6275438/

REFERENCES:
- [Derived] Nantakool S, Reanpang T, Prasannarong M, Pongtam S, Rerkasem K. Upper limb exercise for arteriovenous fistula maturation in people requiring permanent haemodialysis access. Cochrane Database Syst Rev. 2022 Oct 3;10(10):CD013327. doi: 10.1002/14651858.CD013327.pub2. PMID 36184076